CLINICAL TRIAL: NCT06488651
Title: Trajectory of Immunosuppression-Caused Tremor In Kidney and Lung Transplant Recipients
Acronym: TICTIK
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: METc 2022/392; 11036 (Registry Identifier: UMCG Research Registry)
Record Dates: First submitted 2024-06-11; First posted 2024-07-05 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-12

CONDITIONS: Kidney Transplantation; Tremor
Keywords: Kidney transplant recipient; Tremor; Calcineurin inhibitor; Tacrolimus; Cyclosporine
MeSH Terms: conditions — Tremor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Kidney and lung transplant recipients have to adhere to a strict immunosuppressive maintenance regime, generally consisting of calcineurin inhibitors (CNI). Tremor is a common and distressing side effect of CNI-use. To what extent objective and/or subjective tremor changes over time in currently unknown. Therefore, this longitudinal prospective study aimed to assess the course of tremor in the first year after transplantation.

DETAILED DESCRIPTION:
Kidney and lung transplant recipients have to adhere to a strict immunosuppressive maintenance regime, generally including calcineurin inhibitors (CNIs). These CNIs, including cyclosporine and tacrolimus, are essential to prevent graft rejection, but are associated with multiple side-effects. One of the most frequently reported side-effects of CNIs is the development of tremor: rhythmic, sinusoidal oscillations of the limbs, head or trunk. CNI-induced tremor generally occurs soon after initiation of CNI maintenance therapy, and occurs in up to half of kidney transplant recipients who use CNIs. Higher tacrolimus blood concentration has been associated with more severe tremor, and lung transplant recipients have the highest target trough concentration. Thus, tremor may be especially an import symptom for this patient population. To what extent tremor changes over time and whether this change is objective and/or subjective is currently unknown. In-depth investigation of the course of tremor is therefore warranted, which would add valuable information to previous studies on tremor prevalence. We therefore aim to assess the course of tremor in the first year after kidney- and lung transplantation. We expect tremor to become less severe over time after transplantation, because patients CNI dosage decrease with time after transplantation. However, it may also be hypothesized that CNI neurotoxicity may accumulate with consequent worsening of tremor. More information regarding the course of tremor after transplantation is essential to increase understanding of CNI-induced tremor, as well as for patient counselling and future research to alleviate the burden of CNI-induced tremor.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 16 years old, who will receive a kidney transplant or have recieved a kidney or lung transplant

Exclusion Criteria:

* patients who are unable to comprehend the questionnaires and tests

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: hospitalized (future) kidney and lung transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Bain spirographs | From enrollment, before transplantation, to one year after transplantation
  Objective measurement of tremor severity. Spirographs will be assessed blindly by two neurologists, resulting in a score ranging from 0 (best outcome) to 10 (worst outcome) on each spiral.

SECONDARY OUTCOMES:
The visual analog scale (VAS) | From enrollment, before transplantation, to one year after transplantation
  A scale from 0 (no tremor) to 100 (most severe tremor)
Accelerometery | Measurement will be performed for the duration of one day, at a non-specific time-point after transplantation.
  Patients with evident tremor will be invited to briefly (1 minute) wear an wrist accelerometer hourly for one day (9:00-21:00). This accelerometer, which is similar to a watch, allows us to assess tremor variability during the day.
The Fahn-Tolosa-Marin Tremor Rating Scale (FTM-TRS) part B | From enrollment, before transplantation, to one year after transplantation
  The TRS-B relates to action tremors of the upper extremities, particulary writing and pouring liquids. Severity is determined by watching the patient carry out the aforementioned activities, after wich a score is derived that ranges from 0 points (no tremor) to 36 points (most severe tremor).
The Fahn-Tolosa-Marin Tremor Rating Scale (FTM-TRS) part C | From enrollment, before transplantation, to one year after transplantation
  The TRS-C consists of eight questions to assess patient-perceived tremor occurrence during ADL, including writing, speaking, and bringing food or liquids to the mouth. To every question, patients graded the impairment tremor has on ADL with a score ranging from 0 (no influence of tremor on ADL) to 4 (severe influence of tremor on ADL). A total score was calculated by summing the individual scores, with a theoretical minimum score of 0 (no tremor) and a maximum score of 32 points (most severe tremor).

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pirsch JD, Miller J, Deierhoi MH, Vincenti F, Filo RS. A comparison of tacrolimus (FK506) and cyclosporine for immunosuppression after cadaveric renal transplantation. FK506 Kidney Transplant Study Group. Transplantation. 1997 Apr 15;63(7):977-83. doi: 10.1097/00007890-199704150-00013. PMID 9112351
- [Background] David-Neto E, Lemos FBC, Arai Furusawa E, Schwartzman BS, Cavalcante JS, Yagyu EM, Romano P, Ianhez LE. Impact of cyclosporin A pharmacokinetics on the presence of side effects in pediatric renal transplantation. J Am Soc Nephrol. 2000 Feb;11(2):343-349. doi: 10.1681/ASN.V112343. PMID 10665942
- [Background] Erro R, Bacchin R, Magrinelli F, Tomei P, Geroin C, Squintani G, Lupo A, Zaza G, Tinazzi M. Tremor induced by Calcineurin inhibitor immunosuppression: a single-centre observational study in kidney transplanted patients. J Neurol. 2018 Jul;265(7):1676-1683. doi: 10.1007/s00415-018-8904-x. Epub 2018 May 18. PMID 29777361
- [Background] Paul F, Muller J, Christe W, Steinmuller T, Poewe W, Wissel J. Postural hand tremor before and following liver transplantation and immunosuppression with cyclosporine or tacrolimus in patients without clinical signs of hepatic encephalopathy. Clin Transplant. 2004 Aug;18(4):429-33. doi: 10.1111/j.1399-0012.2004.00184.x. PMID 15233821
- [Background] Morgan JC, Kurek JA, Davis JL, Sethi KD. Insights into Pathophysiology from Medication-induced Tremor. Tremor Other Hyperkinet Mov (N Y). 2017 Nov 22;7:442. doi: 10.7916/D8FJ2V9Q. eCollection 2017. PMID 29204312
- [Background] Bhatia KP, Bain P, Bajaj N, Elble RJ, Hallett M, Louis ED, Raethjen J, Stamelou M, Testa CM, Deuschl G; Tremor Task Force of the International Parkinson and Movement Disorder Society. Consensus Statement on the classification of tremors. from the task force on tremor of the International Parkinson and Movement Disorder Society. Mov Disord. 2018 Jan;33(1):75-87. doi: 10.1002/mds.27121. Epub 2017 Nov 30. PMID 29193359
- [Background] Naesens M, Kuypers DR, Sarwal M. Calcineurin inhibitor nephrotoxicity. Clin J Am Soc Nephrol. 2009 Feb;4(2):481-508. doi: 10.2215/CJN.04800908. PMID 19218475
- [Background] Kugler C, Fischer S, Gottlieb J, Tegtbur U, Welte T, Goerler H, Simon A, Haverich A, Strueber M. Symptom experience after lung transplantation: impact on quality of life and adherence. Clin Transplant. 2007 Sep-Oct;21(5):590-6. doi: 10.1111/j.1399-0012.2007.00693.x. PMID 17845632